CLINICAL TRIAL: NCT01446471
Title: REASON 1 Trial: Sonography in Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: North Shore University Hospital (Other); NYU Langone Health (Other); Mount Sinai Hospital, New York (Other); Washington University School of Medicine (Other); University of New Mexico (Other); Wake Forest University Health Sciences (Other); University of California, Irvine (Other); University of Utah (Other); Carolinas Medical Center (Other); Emory University (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Duke University (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Rhode Island Hospital (Other); Christiana Care Health Services (Other); George Washington University (Other); Kingston Health Sciences Centre (Other); University of Ottawa (Other); Jewish General Hospital (Other); Horizon Health Network (Other); York Hospitals (Other); Boston Medical Center (Other); Indiana University (Other); Yale University (Other); Queen's Medical Center (Other); University of Hawaii (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Romolo Gaspari, Director, Division of Emergency Ultrsound, University of Massachusetts, Worcester
Other Study IDs: REASON01
Record Dates: First submitted 2011-09-09; First posted 2011-10-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Cardiac Arrest; Pulseless Electrical Activity; Asystole
Keywords: Bedside Ultrasound; Point of care ultrasound; cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Arrest: Patients in Cardiac Arrest will be enrolled

SUMMARY:
The aim of this study is to investigate the predictive value of the presence or absence of cardiac activity by bedside ultrasound during cardiac arrest. The investigators anticipate based on previous research that patients who suffer a cardiac arrest and have cardiac activity on bedside ultrasound will have a greater chance of surviving to hospital admission. The investigators hypothesis is that the mortality rate in patients in cardiac arrest with no cardiac activity by ultrasound will have a mortality rate of 100%.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational trial involving sites across the United States and Canada. Patients will be enrolled through the emergency department either presenting in cardiac arrest, or going into cardiac arrest while in the emergency department. Patients who develop cardiac arrest as inpatients will also be enrolled at centers capable of enrolling inpatients subjects. Advanced Cardiac Life Support (ACLS) protocols and institutional policies for resuscitation will be followed, as is the current standard of care. A patient encounter will conclude upon halting of cardiopulmonary resuscitation. Final disposition of the patient will be evaluated by chart review.

After the initial cardiac arrest and disposition there will be no further direct patient interactions as part of the study except in the setting of repeat cardiac arrest. Patients that have a repeat arrest can undergo a repeated ultrasound exam if they continue to meet inclusion criteria. The repeat episode will be recorded as a continuation of the event and not as a separate enrollment.

Subject data, with Protected Health Information (PHI) removed, will be uploaded into the REDcap web-based database as soon as possible and within 7 days of final disposition. Data will be obtained from initial patient encounter, patient records, and EMS records when available. Additional data may be obtained by chart review to obtain data points not available at initial contact. Individual sites will keep secured records to enable identification of the patient source if data review is required.

Patient information will include 6 types of data, past medical history, events surrounding the cardiac arrest, actions taken by health care professionals, peri-arrest presentation, peri-arrest interventions, and patient outcomes. Health care professional actions can include ACLS medication administration, airway management, chest compressions, defibrillation, pacing, and other resuscitative interventions. Specific data points are listed in the paper version of electronic Case Report Form, CRF, see Appendix A.

Sonography will not hinder or impair resuscitative efforts in any way, including halting CPR or prolonging pauses in cardiopulmonary rescusitation (CPR). Sonographic images will be obtained during designated pauses in chest compressions, as is routine care, during CPR for pulse checks, rhythm checks, and necessary resuscitative procedures.

Single or multi-view echocardiography will be performed as appropriate to obtain diagnostic information for each particular patient during resuscitative efforts. Recording of the image loops will be performed during image acquisition according to standard technology availability at each site. To facilitate image acquisition, the ultrasound probe may be placed in the epigastrium or parasternal region during CPR with the heart centered in the field of view, if it will not interfere with ongoing resuscitation. Recording of the images can begin immediately upon pauses of CPR using whatever means are available at the site. Sonographic images will be obtained by competent personnel with experience in bedside cardiac ultrasound. This information will be made available to the physician taking care of the patient

Ultrasound images will consist of a single or multiple view(s) that can include subxiphoid, parasternal long axis, and/or apical 4 chamber. While not primarily preferred views; also acceptable are parasternal short axis or apical 2 chamber views. Image requirements will be based on adequate echocardiographic windows and adequate image acquisition as determined by the physician performing the bedside ultrasound. In the setting of difficult to image patients a combination of views may be required to obtain adequate information.

There will be at least two ultrasound exams performed. The initial ultrasound exam and video will be obtained upon the first pause for pulse or rhythm check once the inclusion criteria are met and no exclusion criteria are present. The final ultrasound exam and video will be obtained when resuscitative efforts are halted.

All ultrasound images will be recorded for later review by the Regional Coordinating Site for each Local Site. Ultrasound videos will be interpreted during acquisition as cardiac activity present or absent and valvular movement present or absent. Specific video file formats that are acceptable include MPEG4, Quicktime (MOV), DV, AVI, and WMV. Files will be forwarded at least monthly to the Site Coordinator for the Regional Site and sent within 1 week of request by the regional coordinating site.

INITIAL INTERPRETATION OF CARDIAC IMAGES The Local Site PI will interpret ultrasound images and the information will be uploaded into the central database or another database specified by the Central Coordinating Site. Cardiac activity will initially categorize as "Cardiac Activity Present", "Cardiac Activity Absent", Valve Movement Present", or Valve Movement Absent". Cardiac activity is defined as any intrinsic movement of the myocardium, but not isolated movement of the cardiac valves. Valve movement is defined as any movement of the cardiac valves.

FINAL INTERPRETATION OF CARDIAC IMAGES

Cardiac images will be reviewed by regional site PIs for sub-categories of cardiac activity. A heart with any intrinsic cardiac movement outside of isolated valvular motion will be categorized as "Cardiac Activity Present". Ultrasound images in patients with cardiac activity will be further categorized as:

1. Cardiac motion but No decrease in chamber size
2. Cardiac motion with a decrease in chamber size <10%
3. Cardiac motion with a decrease in chamber size of >10%.

The estimated duration that each subject will participate is the length of the cardiopulmonary resuscitation which can vary by patient, but can be from 15 minutes to 1 hour, with later follow up (hours to days later) to determine final disposition.

A summary of the sequence and duration of all research activities is as follows.

Patient interactions (estimated 15 minutes to 1 hour)

* Patient identified to be in cardiac arrest with confirmation of no pulse.
* Chest compressions and ACLS protocols initiated as per standard care
* Bedside ultrasound of heart performed and interpreted during standard pauses in cardiac compressions as per routine care at institution (3-6 seconds)
* ACLS protocols continue as per standard care by treating physician
* Resuscitation activities halted by either pronouncement of patient or return of spontaneous circulation allowing disposition planning
* Bedside ultrasound of heart performed and interpreted (3-6 seconds)

Data Acquisition (Immediate to days later via chart review)

* Final patient disposition determined
* Interval events recorded (ie: repeat cardiopulmonary arrest)

Data Management (immediate to days or weeks later)

* Subject data with PHI removed entered into research database
* Subject data with PHI removed updated in research database if CRF not completed initially
* Cardiac ultrasound images with PHI removed sent to regional site for review

ELIGIBILITY:
Inclusion Criteria:

* Patients in cardiac arrest with no pulse

Exclusion Criteria:

* Patients with isolated ventricular fibrillation as their cardiac rhythm at the time of presentation
* Traumatic cardiopulmonary arrest
* Ultrasound system or physician experienced in bedside cardiac ultrasound not available
* Resuscitative efforts halted due to end of life decisions or designations
* Attending physician of record declines enrollment of patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2010-01; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of patients that survive to Hospital Discharge | Up to 12 months
  Participants will be followed for the duration of hospital stay, an expected average of up to 12 months. The time frame is an estimate based on previous research. Patients could survive hours to days to weeks or months.

SECONDARY OUTCOMES:
The number of patients that demonstrate a Return of Spontaneous Circulation | Up to 60 Minutes -
  Participants will be followed until a demonstrated return of spontaneous circulation (i.e. regain a pulse and blood pressure) is present - an expected average of up to 60 minutes. The time frame is an estimate based on previous research but is in the order of minutes.
The number of patients that survive to hospital admission | Up to 24 hours
  Surviving participants will be followed to hospital admission- an expected average of up to 24 hours. The time frame is an estimate based on previous research. Patients could survive minutes to hours before they are admitted.

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD, PhD, Principal Investigator — UMass Memorial Health
Locations (7):
- United States (6):
  - Christiana Health Care, Newark, Delaware
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Washington University Hospital, St Louis, Missouri
  - Northshore University Hospital, Manhasset, New York
  - Carolinas Medical Center, Charlotte, North Carolina
- University of Ottowa, Ottowa, Canada